CLINICAL TRIAL: NCT05347147
Title: A Phase III Randomised, Placebo-controlled, Double-blind, Multi-centre, Clinical Trial to Determine the Efficacy and Safety of Presendin in Idiopathic Intracranial Hypertension
Brief Title: A Trial to Determine the Efficacy and Safety of Presendin in IIH
Acronym: IIH EVOLVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Following a strategic evaluation of its IIH EVOLVE Phase III clinical trial investigating Presendin™, the Invex Board has made the difficult decision that the continuation of the trial is not viable and therefore the trial has been terminated.
Sponsor: Invex Therapeutics Ltd. (Industry)
Collaborators: Premier Research (Other); University Hospital Birmingham (Other); University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INVEX-CLIN-IIH-301
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Idiopathic Intracranial Hypertension
Keywords: Presendin
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Intervention Model Description: This will be a placebo-controlled, double-blind, multi-centre clinical trial in approximately 240 randomised patients with IIH.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators and other site personnel, patients, contract research organisation and Sponsor personnel will be blinded regarding the treatment during the randomised period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Presendin (Experimental): 2.0 mg
  Interventions: Drug: Presendin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Presendin — Presendin is supplied as 2 parts, one vial consisting of a drug part (white or greyish white powder in a clear vial) and one pre-filled syringe containing the diluent part (colourless liquid). The drug part is suspended in the diluent part solution and administered SC as a suspension.
  Arms: Presendin
Drug: Placebo — Placebo is supplied as 2 parts (visually identical to the Presendin vial and pre-filled diluent syringe). The drug part will exclude the active pharmaceutical ingredient (exenatide acetate) and the diluent part will be the same as the active treatment diluent. The drug part is suspended in the diluent part solution and administered SC as a suspension.
  Arms: Placebo

SUMMARY:
Idiopathic intracranial hypertension (IIH) has significant associated morbidity and reduced quality of life. There is a significant risk of visual loss and patients also typically suffer with chronic disabling headaches.

This trial has been designed to evaluate the efficacy and safety of a new formulation of exenatide (Presendin) in the reduction of intracranial pressure (ICP) in patients with IIH.

DETAILED DESCRIPTION:
Patients will be provided with training on the self-administration of the trial medication from the site trial co-ordinator.

A 1-week screening period will be followed by a 24-week randomised double-blind treatment period in which patients will be randomised (1:1) to receive a subcutaneous (SC) dose of either Presendin (containing 2 mg of exenatide [active group]) or matching placebo (placebo group), self-administered once weekly.

At the end of the randomised treatment period (Week 24), all patients will have an end-of-treatment clinic visit. Five weeks after the end-of-treatment visit, an end-of-trial safety follow-up telephone visit will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of consent.
2. Diagnosis of new IIH by consensus criteria, including normal structural brain imaging (excluding features of raised ICP and incidentalomas), including either magnetic resonance venography or computed tomographic venography to exclude thrombosis and no evidence of a secondary causes of raised ICP.
3. Newly diagnosed patients with screening commenced no more than 4 weeks after the diagnostic LP.
4. Lumbar puncture opening pressure ≥25 cm cerebrospinal fluid (CSF) at diagnosis.
5. Presence of bilateral papilloedema (Frisén grade ≥1). Verification of papilloedema by the OCT Reading Centre. Where there is uncertainty fundus photography and/or ultrasound scan (B scan) of the optic nerves should be conducted for evaluation by the Independent Adjudication Committee (IAC).
6. Perimetric Mean Deviation defined as between -2 to -7 decibels (dB) in at least one eye. Eyes meeting this criterion will defined as 'study eyes'.
7. Reproducible visual loss present on automated perimetry including no more than 15% false positive responses (reliability confirmed by the Visual Field Reading Centre) in study eyes.
8. Two or more headache days over the 7-day period prior to screening and also the patient must meet this criterion during the 7-day screening period.
9. Females of childbearing potential must have a negative pregnancy test and must agree to use a highly effective birth control method (failure rate less than 1% per year when used consistently and correctly) during the whole trial duration including the last follow-up visit (12 weeks after ceasing drug). Female patients who are lactating must agree to stop breast-feeding OR Female patients of non-childbearing potential (defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or post-menopausal females defined as 12 months of amenorrhoea [in questionable cases a blood sample with simultaneous follicle stimulation hormone 25-140 IE/L and oestradiol <200 pmol/L is confirmatory]).
10. Male patients with a female partner of childbearing potential must commit to practice methods of contraception (e.g., condom, vasectomy) and abstain from sperm donation during the trial including the last follow-up visit (12 weeks after ceasing drug). Their partners, if they are women of childbearing potential, must agree to practice contraception and to use a highly effective method of contraception during the trial, including the last follow-up visit (12 weeks after ceasing drug).
11. Able to provide written informed consent.

Exclusion Criteria:

IIH-related exclusion criteria:

1. Presence of venous sinus thrombosis on brain imaging by either magnetic resonance or computerised tomographic venography.
2. Previous IIH surgery including CSF shunt, optic nerve sheath fenestration or dural venous sinus stent or sub-temporal decompression.
3. Previous bariatric surgery within the last 3 months or intention during the trial.
4. Abnormal neurological examination (aside from papilloedema and consequent visual loss or sixth or seventh nerve palsy or palsies).
5. Treatment to lower ICP within 1 week prior to screening visit (e.g., acetazolamide, topiramate [including if used as a migraine preventative], diuretics, glucocorticoids [I.V., injectable steroids or oral (including dexamethasone and prednisolone)]). Nasal, inhaled, or topical steroids are allowed.
6. Use of any drugs known to cause intracranial hypertension, including exposure to fluoroquinolones, lithium, vitamin A, or tetracyclines within 2 months prior to diagnostic LP.

   Vision-related exclusion criteria:
7. Any disease other than refractive error that causes visual loss in the study eyes. Where there is uncertainty this would be determined by the IAC.
8. Refractive error worse than +/- 6.00 sphere or worse than +/- 3.00 cylinder in study eyes. In addition, participants with myopia of worse than -6.00 D sphere but less than or equal to -8.00 D sphere are eligible if the subject wears a contact lens for all perimetry examinations with the appropriate correction.
9. Inability to perform a reliable visual field examination as deemed by the Visual Field Reading Centre in the study eyes. Where there is uncertainty this would be evaluated by the IAC.

   Headache-related exclusion criteria:
10. Does not complete ≥6 days of electronic/paper trial diary during the 7-day screening period.

    Other exclusion criteria:
11. Untreated previously diagnosed obstructive sleep apnoea with historically recorded apnoea-hypopnea index greater than 15.
12. Glucagon like peptide-1 receptor agonist within last 4 weeks prior to screening.
13. COVID-19 vaccine within 2 weeks prior to screening.
14. Allergy/known hypersensitivity to the active substance and/or excipients of the investigational product.
15. Has known contraindications to glucagon like peptide-1 (GLP-1) receptor agonists (e.g., ketoacidosis, severe gastrointestinal disease, pancreatitis, renal impairment) which may affect the safety of the patient.
16. Using any glucose-lowering medication.
17. Currently taking warfarin.
18. Alanine transaminase (ALT) or aspartate transaminase (AST) ≥2x the upper limit of normal (ULN), total bilirubin ≥1.5x ULN, or alkaline phosphatase (ALP) ≥1.5 ULN at screening. Note - patients with elevated total bilirubin are not excluded if they meet criteria for Gilbert's syndrome, including: bilirubin is predominantly indirect (with normal direct bilirubin level); and ALT, AST and ALP ≤1x ULN).
19. Kidney disease (as defined by serum cystatin C-based estimated glomerular filtration rate <55 mL/min/1.73 m², calculated at investigator site).
20. Any of the following abnormalities in clinical laboratory tests at screening, as assessed by the central laboratory and confirmed by a single repeat, if deemed necessary: Haemoglobin <10 g/dL (<100 g/L); Platelet count <75 x 10⁹/L (<75,000/mm³).
21. Using recreational or illicit drugs at the time of signing the informed consent, or recent history (within the last year) of drug or alcohol abuse or dependence according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition criteria, that in the opinion of the investigator puts the patient at risk.
22. Is unable to self-administer the trial medication (or unable to administer trial medication with support) after receiving training during the screening period.
23. History of any clinically significant disease or disorder that, in the opinion of the investigator, may either put the patient at risk because of participation in the trial or influence the results or the patient's ability to participate in the trial.
24. Any contraindication to lumbar puncture procedure in the opinion of the investigator.
25. Has participated in any other interventional trial within 1 month prior to the screening visit.
26. Is pregnant or breastfeeding.

Note: Use of headache preventative medication is allowed at enrolment (except for topiramate). Changes to headache preventative medication during the trial should be made in consultation with the IAC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (7):
  - UCHealth Sue Anschutz-Rodgers Eye Center - Anschutz Medical Campus, Aurora, Colorado
  - University of Miami Leonard M. Miller School of Medicine (UMMSM) - Bascom Palmer Eye Institute, Miami, Florida
  - University of Minnesota Health, Minneapolis, Minnesota
  - New York Eye and Ear Infirmary of Mount Sinai, New York, New York
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Neuro-Eye Clinical Trials, Inc, Houston, Texas
- Australia (4):
  - Liverpool Hospital, Liverpool, New South Wales
  - Sydney Eye Hospital, Sydney, New South Wales
  - Vision SA, Kent Town, South Australia
  - Alfred Health - The Alfred Centre, Melbourne, Victoria
- Germany (4):
  - University Hospital Bonn, Bonn
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsmedizin Mainz, Mainz
  - University Hospital Muenster, Department Ophthalmology Clinical Trials in Ophthalmology (CTO), Münster
- Israel (6):
  - Rambam Medical Center, Haifa
  - Bnai Zion Medical Center, Haifa
  - The Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center - Ein Karem, Jerusalem
  - Pade Medical Center (Poriya), Tiberias
- New Zealand Clinical Research (Aukland), Auckland, New Zealand
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust - Queen Elizabeth Hospital Birmingham, Birmingham
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Presendin | Placebo
Started | 8 | 6
Completed | 3 | 1
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Sponsor request | 3 | 3
Not completed — Study termination | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Presendin | Placebo | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.0 (8.5) | 28.5 (5.32) | 28.2 (7.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 7 | 3 | 10
  More than 1 Race | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 3 | 1 | 4
  United States | 1 | 0 | 1
  United Kingdom | 0 | 1 | 1
  Australia | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in ICP From Baseline to Week 24 Measured by Lumbar Puncture (LP), Where a Higher LP Value Indicates Greater ICP
Description: ICP was measured by LP (opening pressure) using an LP manometer; Baseline and Week 24 ICP values (measured in cm CSF) are presented for each subject. A standard operating procedure was followed by all study sites for all study-related ICP measurements by LP.
Time Frame: Baseline to Week 24
Population: Data presented represents collected data from individual subjects. For subject anonymity, study-assigned subject IDs are not included here, and subject numbers used throughout the ClinicalTrials.gov results do not consistently relate to the same subjects.
Measure: Number; unit: cm CSF
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 2 | 1
cm CSF
  Subject 1 Baseline ICP: number analyzed (Participants) | 1 | 0
  Subject 1 Baseline ICP | 25 |
  Subject 1 Week 24 ICP: number analyzed (Participants) | 1 | 0
  Subject 1 Week 24 ICP | 28 |
  Subject 2 Baseline ICP: number analyzed (Participants) | 1 | 0
  Subject 2 Baseline ICP | 28 |
  Subject 2 Week 24 ICP: number analyzed (Participants) | 1 | 0
  Subject 2 Week 24 ICP | 29 |
  Subject 3 Baseline ICP: number analyzed (Participants) | 0 | 1
  Subject 3 Baseline ICP |  | 40
  Subject 3 Week 24 ICP: number analyzed (Participants) | 0 | 1
  Subject 3 Week 24 ICP |  | 30

2. Secondary Outcome: Change in Perimetric Mean Deviation (PMD), Measured by Humphrey Visual Field (HVF) Analysis (24-2 SITA-Standard), Where a Larger Negative Result Indicates Greater Visual Loss
Time Frame: Baseline to Week 24
Population: Data presented represent collected data from individual subjects for study eyes only. Baseline PMD had to be -2 dB to -7 dB for an eye to count as a "study eye". For subject anonymity, study-assigned subject IDs are not included here, and subject numbers used throughout the ClinicalTrials.gov results do not consistently relate to the same subjects.
Measure: Number; unit: dB
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 4 | 5
dB
  Subject 1: right eye, Baseline PMD: number analyzed (Participants) | 1 | 0
  Subject 1: right eye, Baseline PMD | -5.89 |
  Subject 1: right eye, Week 24 PMD: number analyzed (Participants) | 1 | 0
  Subject 1: right eye, Week 24 PMD | 0.74 |
  Subject 2: right eye, Baseline PMD: number analyzed (Participants) | 1 | 0
  Subject 2: right eye, Baseline PMD | -3.60 |
  Subject 2: right eye, Week 24 PMD: number analyzed (Participants) | 1 | 0
  Subject 2: right eye, Week 24 PMD | -1.09 |
  Subject 3: right eye, Baseline PMD: number analyzed (Participants) | 0 | 1
  Subject 3: right eye, Baseline PMD |  | -2.79
  Subject 3: right eye, Week 24 PMD: number analyzed (Participants) | 0 | 1
  Subject 3: right eye, Week 24 PMD |  | -1.50
  Subject 3: left eye, Baseline PMD: number analyzed (Participants) | 0 | 1
  Subject 3: left eye, Baseline PMD |  | -4.78
  Subject 3: left eye, Week 24 PMD: number analyzed (Participants) | 0 | 1
  Subject 3: left eye, Week 24 PMD |  | -2.33
  Subject 4: right eye, Baseline PMD: number analyzed (Participants) | 0 | 1
  Subject 4: right eye, Baseline PMD |  | -3.16
  Subject 4: right eye, Week 24 PMD: number analyzed (Participants) | 0 | 1
  Subject 4: right eye, Week 24 PMD |  | -2.20
  Subject 4: left eye, Baseline PMD: number analyzed (Participants) | 0 | 1
  Subject 4: left eye, Baseline PMD |  | -2.36
  Subject 4: left eye, Week 24 PMD: number analyzed (Participants) | 0 | 1
  Subject 4: left eye, Week 24 PMD |  | -1.60
  Subject 5: right eye, Baseline PMD: number analyzed (Participants) | 0 | 1
  Subject 5: right eye, Baseline PMD |  | -2.24
  Subject 5: right eye, Week 24 PMD: number analyzed (Participants) | 0 | 1
  Subject 5: right eye, Week 24 PMD |  | -2.69
  Subject 5: left eye, Baseline PMD: number analyzed (Participants) | 0 | 1
  Subject 5: left eye, Baseline PMD |  | -3.66
  Subject 5: left eye, Week 24 PMD: number analyzed (Participants) | 0 | 1
  Subject 5: left eye, Week 24 PMD |  | -2.98
  Subject 6: right eye, Baseline PMD: number analyzed (Participants) | 1 | 0
  Subject 6: right eye, Baseline PMD | -3.64 |
  Subject 6: right eye, Week 24 PMD: number analyzed (Participants) | 1 | 0
  Subject 6: right eye, Week 24 PMD | -0.88 |
  Subject 6: left eye, Baseline PMD: number analyzed (Participants) | 1 | 0
  Subject 6: left eye, Baseline PMD | -2.55 |
  Subject 6: left eye, Week 24 PMD: number analyzed (Participants) | 1 | 0
  Subject 6: left eye, Week 24 PMD | 0.15 |
  Subject 7: right eye, Baseline PMD: number analyzed (Participants) | 0 | 1
  Subject 7: right eye, Baseline PMD |  | -2.54
  Subject 7: right eye, Week 24 PMD: number analyzed (Participants) | 0 | 1
  Subject 7: right eye, Week 24 PMD |  | -0.49
  Subject 7: left eye, Baseline PMD: number analyzed (Participants) | 0 | 1
  Subject 7: left eye, Baseline PMD |  | -3.15
  Subject 7: left eye, Week 24 PMD: number analyzed (Participants) | 0 | 1
  Subject 7: left eye, Week 24 PMD |  | -0.26
  Subject 8: left eye, Baseline PMD: number analyzed (Participants) | 0 | 1
  Subject 8: left eye, Baseline PMD |  | -2.6
  Subject 8: left eye, Week 24 PMD: number analyzed (Participants) | 0 | 1
  Subject 8: left eye, Week 24 PMD |  | -1.5
  Subject 9: right eye, Baseline PMD: number analyzed (Participants) | 1 | 0
  Subject 9: right eye, Baseline PMD | -2.37 |
  Subject 9: right eye, Week 24 PMD: number analyzed (Participants) | 1 | 0
  Subject 9: right eye, Week 24 PMD | -2.59 |
  Subject 9: left eye, Baseline PMD: number analyzed (Participants) | 1 | 0
  Subject 9: left eye, Baseline PMD | -3.81 |
  Subject 9: left eye, Week 24 PMD: number analyzed (Participants) | 1 | 0
  Subject 9: left eye, Week 24 PMD | -2.04 |

3. Secondary Outcome: Papilloedema by Change in Retinal Nerve Fibre Layer (RNFL) Thickness, With a Greater Thickness of RNFL Indicating Greater Swelling and Greater Extent of Papilloedema
Time Frame: Baseline to Week 24
Population: Data presented represents collected data from individual subjects for study eyes only. Baseline PMD had to be -2 dB to -7 dB for an eye to count as a "study eye". For subject anonymity, study-assigned subject IDs are not included here, and subject numbers used throughout the ClinicalTrials.gov results do not consistently relate to the same subjects. Cirrus was the imaging platform used for all subjects except Subjects 6 and 7, where Zeiss was used.
Measure: Number; unit: µm
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 4 | 4
µm
  Subject 1: right eye, Baseline RNFL: number analyzed (Participants) | 1 | 0
  Subject 1: right eye, Baseline RNFL | 115 |
  Subject 1: right eye, Week 24 RNFL: number analyzed (Participants) | 1 | 0
  Subject 1: right eye, Week 24 RNFL | 105 |
  Subject 2: right eye, Baseline RNFL: number analyzed (Participants) | 1 | 0
  Subject 2: right eye, Baseline RNFL | 199 |
  Subject 2: right eye, Week 24 RNFL: number analyzed (Participants) | 1 | 0
  Subject 2: right eye, Week 24 RNFL | 173 |
  Subject 3: right eye, Baseline RNFL: number analyzed (Participants) | 0 | 1
  Subject 3: right eye, Baseline RNFL |  | 140
  Subject 3: right eye, Week 24 RNFL: number analyzed (Participants) | 0 | 1
  Subject 3: right eye, Week 24 RNFL |  | 155
  Subject 3: left eye, Baseline RNFL: number analyzed (Participants) | 0 | 1
  Subject 3: left eye, Baseline RNFL |  | 114
  Subject 3: left eye, Week 24 RNFL: number analyzed (Participants) | 0 | 1
  Subject 3: left eye, Week 24 RNFL |  | 122
  Subject 4: right eye, Baseline RNFL: number analyzed (Participants) | 0 | 1
  Subject 4: right eye, Baseline RNFL |  | 432
  Subject 4: right eye, Week 24 RNFL: number analyzed (Participants) | 0 | 1
  Subject 4: right eye, Week 24 RNFL |  | 372
  Subject 4: left eye, Baseline RNFL: number analyzed (Participants) | 0 | 1
  Subject 4: left eye, Baseline RNFL |  | 358
  Subject 4: left eye, Week 24 RNFL: number analyzed (Participants) | 0 | 1
  Subject 4: left eye, Week 24 RNFL |  | 317
  Subject 5: right eye, Baseline RNFL: number analyzed (Participants) | 0 | 1
  Subject 5: right eye, Baseline RNFL |  | 127
  Subject 5: right eye, Week 24 RNFL: number analyzed (Participants) | 0 | 1
  Subject 5: right eye, Week 24 RNFL |  | 119
  Subject 5: left eye, Baseline RNFL: number analyzed (Participants) | 0 | 1
  Subject 5: left eye, Baseline RNFL |  | 121
  Subject 5: left eye, Week 24 RNFL: number analyzed (Participants) | 0 | 1
  Subject 5: left eye, Week 24 RNFL |  | 126
  Subject 6: right eye, Baseline RNFL: number analyzed (Participants) | 1 | 0
  Subject 6: right eye, Baseline RNFL | 111 |
  Subject 6: right eye, Week 24 RNFL: number analyzed (Participants) | 1 | 0
  Subject 6: right eye, Week 24 RNFL | 101 |
  Subject 6: left eye, Baseline RNFL: number analyzed (Participants) | 1 | 0
  Subject 6: left eye, Baseline RNFL | 111 |
  Subject 6: left eye, Week 24 RNFL: number analyzed (Participants) | 1 | 0
  Subject 6: left eye, Week 24 RNFL | 105 |
  Subject 7: right eye, Baseline RNFL: number analyzed (Participants) | 0 | 1
  Subject 7: right eye, Baseline RNFL |  | 114
  Subject 7: right eye, Week 24 RNFL: number analyzed (Participants) | 0 | 1
  Subject 7: right eye, Week 24 RNFL |  | 107
  Subject 7: left eye, Baseline RNFL: number analyzed (Participants) | 0 | 1
  Subject 7: left eye, Baseline RNFL |  | 119
  Subject 7: left eye, Week 24 RNFL: number analyzed (Participants) | 0 | 1
  Subject 7: left eye, Week 24 RNFL |  | 111
  Subject 8: right eye, Baseline RNFL: number analyzed (Participants) | 1 | 0
  Subject 8: right eye, Baseline RNFL | 81 |
  Subject 8: right eye, Week 24 RNFL: number analyzed (Participants) | 1 | 0
  Subject 8: right eye, Week 24 RNFL | 74 |
  Subject 8: left eye, Baseline RNFL: number analyzed (Participants) | 1 | 0
  Subject 8: left eye, Baseline RNFL | 132 |
  Subject 8: left eye, Week 24 RNFL: number analyzed (Participants) | 1 | 0
  Subject 8: left eye, Week 24 RNFL | 92 |

4. Secondary Outcome: Papilloedema by Percent Change in Optic Nerve Head Size, Measured by Optical Coherence Tomography (OCT), Where a Larger Optic Nerve Head Size Reflects Greater Swelling and a Greater Extent of Papilloedema
Time Frame: Baseline to Week 24
Population: Data presented represents collected data from individual subjects for study eyes only. Baseline PMD had to be -2 dB to -7 dB for an eye to count as a "study eye". For subject anonymity, study-assigned subject IDs are not included here, and subject numbers used throughout the ClinicalTrials.gov results do not consistently relate to the same subjects.
Measure: Number; unit: percentage change
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 3 | 4
percentage change
  Subject 1, right eye: number analyzed (Participants) | 1 | 0
  Subject 1, right eye | -6.67 |
  Subject 2, right eye: number analyzed (Participants) | 1 | 0
  Subject 2, right eye | 18.64 |
  Subject 3, right eye: number analyzed (Participants) | 0 | 1
  Subject 3, right eye |  | 8.61
  Subject 3, left eye: number analyzed (Participants) | 0 | 1
  Subject 3, left eye |  | 2.61
  Subject 4, right eye: number analyzed (Participants) | 0 | 1
  Subject 4, right eye |  | 0.77
  Subject 4, left eye: number analyzed (Participants) | 0 | 1
  Subject 4, left eye |  | 2.35
  Subject 5, right eye: number analyzed (Participants) | 0 | 1
  Subject 5, right eye |  | -1.53
  Subject 5, left eye: number analyzed (Participants) | 0 | 1
  Subject 5, left eye |  | 11.41
  Subject 6, right eye: number analyzed (Participants) | 1 | 0
  Subject 6, right eye | -11.87 |
  Subject 6, left eye: number analyzed (Participants) | 1 | 0
  Subject 6, left eye | -8.10 |
  Subject 7, right eye: number analyzed (Participants) | 0 | 1
  Subject 7, right eye |  | -2.82
  Subject 7, left eye: number analyzed (Participants) | 0 | 1
  Subject 7, left eye |  | -6.46

5. Secondary Outcome: The Number of Monthly Headache Days (MHD)
Description: Monthly headache days (according to daily headache diary) = number of days recorded in a 28-day window where data were collected on >7 days and where ≥1 headache on a day met the following criteria:
  * Onset, continuation, or recurrence of headache
  * Any severity or phenotype of headache
  * Lasts at least 30 minutes
  Baseline headache frequency was calculated over the 7 days prior to the randomization visit; ≥5 days of headache data were needed to obtain a valid baseline value. The number of headache days recorded for a period were linearly scaled by the total number of days of data collected in the period for each subject to give the MHD during the baseline period (linearly scaled to a maximum of 28 days) and the last 28-day period during which data were collected on >7 days for each subject prior to study completion or discontinuation.
  Period 1 = Weeks 1-4 Period 2 = Weeks 5-8 Period 3 = Weeks 9-12 Period 4 = Weeks 13-16 Period 5 = Weeks 17-20 Period 6 = Weeks 21-24
Time Frame: Baseline to Week 24
Population: Data presented represents collected data from individual subjects. For subject anonymity, study-assigned subject IDs are not included here, and subject numbers used throughout the ClinicalTrials.gov results do not consistently relate to the same subjects.
  The number of days on which data were collected for each subject during the 7-day baseline period and the last 28-day period are provided in parentheses in the row titles.
  No data were collected for Subject 7 during the 7-day baseline period.
Measure: Number; unit: Monthly headache days
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 8 | 6
Monthly headache days
  Subject 1 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 1 Baseline (5 days) | 28 |
  Subject 1 28-day period 6 (14 days): number analyzed (Participants) | 1 | 0
  Subject 1 28-day period 6 (14 days) | 28 |
  Subject 2 Baseline (7 days): number analyzed (Participants) | 1 | 0
  Subject 2 Baseline (7 days) | 20 |
  Subject 2 28-day period 6 (24 days): number analyzed (Participants) | 1 | 0
  Subject 2 28-day period 6 (24 days) | 3.5 |
  Subject 3 Baseline (7 days): number analyzed (Participants) | 0 | 1
  Subject 3 Baseline (7 days) |  | 28
  Subject 3 28-day period 6 (9 days): number analyzed (Participants) | 0 | 1
  Subject 3 28-day period 6 (9 days) |  | 28
  Subject 4 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 4 Baseline (5 days) | 28 |
  Subject 4 28-day period 4 (11 days): number analyzed (Participants) | 1 | 0
  Subject 4 28-day period 4 (11 days) | 28 |
  Subject 5 Baseline (2 days): number analyzed (Participants) | 1 | 0
  Subject 5 Baseline (2 days) | NA — Data were collected on 2 days, therefore the baseline value was not valid |
  Subject 5 28-day period 4 (10 days): number analyzed (Participants) | 1 | 0
  Subject 5 28-day period 4 (10 days) | 5.6 |
  Subject 6 Baseline (4 days): number analyzed (Participants) | 0 | 1
  Subject 6 Baseline (4 days) |  | NA — Data were collected on 4 days, therefore the baseline value was not valid
  Subject 6 28-day period 2 (10 days): number analyzed (Participants) | 0 | 1
  Subject 6 28-day period 2 (10 days) |  | 11.2
  Subject 7 Baseline (0 days): number analyzed (Participants) | 0 | 0
  Subject 7 28-day period 4 (7 days): number analyzed (Participants) | 0 | 1
  Subject 7 28-day period 4 (7 days) |  | 16
  Subject 8 Baseline (6 days): number analyzed (Participants) | 0 | 1
  Subject 8 Baseline (6 days) |  | 23.33
  Subject 8 28-day period 2 (8 days): number analyzed (Participants) | 0 | 1
  Subject 8 28-day period 2 (8 days) |  | 28
  Subject 9 Baseline (6 days): number analyzed (Participants) | 1 | 0
  Subject 9 Baseline (6 days) | 14 |
  Subject 9 28-day period 6 (18 days): number analyzed (Participants) | 1 | 0
  Subject 9 28-day period 6 (18 days) | 9.33 |
  Subject 10 Baseline (7 days): number analyzed (Participants) | 1 | 0
  Subject 10 Baseline (7 days) | 20 |
  Subject 10 28-day period 4 (12 days): number analyzed (Participants) | 1 | 0
  Subject 10 28-day period 4 (12 days) | 18.67 |
  Subject 11 Baseline (7 days): number analyzed (Participants) | 0 | 1
  Subject 11 Baseline (7 days) |  | 20
  Subject 11 28-day period 4 (15 days): number analyzed (Participants) | 0 | 1
  Subject 11 28-day period 4 (15 days) |  | 5.6
  Subject 12 Baseline (4 days): number analyzed (Participants) | 1 | 0
  Subject 12 Baseline (4 days) | NA — Data were collected on 4 days, therefore the baseline value was not valid |
  Subject 12 28-day period 1(27 days): number analyzed (Participants) | 1 | 0
  Subject 12 28-day period 1(27 days) | 23.85 |
  Subject 13 Baseline (7 days): number analyzed (Participants) | 0 | 1
  Subject 13 Baseline (7 days) |  | 20
  Subject 13 28-day period 4 (21 days): number analyzed (Participants) | 0 | 1
  Subject 13 28-day period 4 (21 days) |  | 1.3
  Subject 14 Baseline (3 days): number analyzed (Participants) | 1 | 0
  Subject 14 Baseline (3 days) | NA — Data were collected on 3 days, therefore the baseline value was not valid |
  Subject 14 28-day period 3 (10 days): number analyzed (Participants) | 1 | 0
  Subject 14 28-day period 3 (10 days) | 0 |

6. Secondary Outcome: Number of Moderate to Severe MHD
Description: Moderate to severe (m-s) MHD (according to daily headache diary) = number of days recorded in a 28-day window where data were collected on >7 days and where ≥1 headache on a day met the following criteria:
  * Severity was of moderate or severe pain and lasted at least 4 hours or,
  * Required acute headache analgesics
  Baseline m-s headache frequency was calculated over the 7 days prior to the randomization visit; ≥5 days of headache data were needed to obtain a valid baseline value. The number of m-s headache days recorded for a period were linearly scaled by the total number of days of data collected in the period for each subject to give the m-s MHD during the baseline period (linearly scaled to a max 28 days) and the last 28-day period during which data were collected on >7 days for each subject prior to study completion or discontinuation.
  Period 1 = Weeks 1-4 Period 2 = Weeks 5-8 Period 3 = Weeks 9-12 Period 4 = Weeks 13-16 Period 5 = Weeks 17-20 Period 6 = Weeks 21-24
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Number; unit: Monthly headache days
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 8 | 6
Monthly headache days
  Subject 1 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 1 Baseline (5 days) | 5.6 |
  Subject 1 28-day period 6 (14 days): number analyzed (Participants) | 1 | 0
  Subject 1 28-day period 6 (14 days) | 10 |
  Subject 2 Baseline (7 days): number analyzed (Participants) | 1 | 0
  Subject 2 Baseline (7 days) | 12 |
  Subject 2 28-day period 6 (24 days): number analyzed (Participants) | 1 | 0
  Subject 2 28-day period 6 (24 days) | 1.167 |
  Subject 3 Baseline (7 days): number analyzed (Participants) | 0 | 1
  Subject 3 Baseline (7 days) |  | 8
  Subject 3 28-day period 6 (9 days): number analyzed (Participants) | 0 | 1
  Subject 3 28-day period 6 (9 days) |  | 24.889
  Subject 4 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 4 Baseline (5 days) | 16.8 |
  Subject 4 28-day period 4 (11 days): number analyzed (Participants) | 1 | 0
  Subject 4 28-day period 4 (11 days) | 28 |
  Subject 5 Baseline (2 days): number analyzed (Participants) | 1 | 0
  Subject 5 Baseline (2 days) | NA — Data were collected on 2 days, therefore the baseline value was not valid |
  Subject 5 28-day period 4 (10 days): number analyzed (Participants) | 1 | 0
  Subject 5 28-day period 4 (10 days) | 0 |
  Subject 6 Baseline (4 days): number analyzed (Participants) | 0 | 1
  Subject 6 Baseline (4 days) |  | NA — Data were collected on 4 days, therefore the baseline value was not valid
  Subject 6 28-day period 2 (10 days): number analyzed (Participants) | 0 | 1
  Subject 6 28-day period 2 (10 days) |  | 5.6
  Subject 7 Baseline (0 days): number analyzed (Participants) | 0 | 0
  Subject 7 28-day period 4 (7 days): number analyzed (Participants) | 0 | 1
  Subject 7 28-day period 4 (7 days) |  | 0
  Subject 8 Baseline (6 days): number analyzed (Participants) | 0 | 1
  Subject 8 Baseline (6 days) |  | 9.333
  Subject 8 28-day period 2 (8 days): number analyzed (Participants) | 0 | 1
  Subject 8 28-day period 2 (8 days) |  | 28
  Subject 9 Baseline (6 days): number analyzed (Participants) | 1 | 0
  Subject 9 Baseline (6 days) | 14 |
  Subject 9 28-day period 6 (18 days): number analyzed (Participants) | 1 | 0
  Subject 9 28-day period 6 (18 days) | 0 |
  Subject 10 Baseline (7 days): number analyzed (Participants) | 1 | 0
  Subject 10 Baseline (7 days) | 20 |
  Subject 10 28-day period 4 (12 days): number analyzed (Participants) | 1 | 0
  Subject 10 28-day period 4 (12 days) | 14 |
  Subject 11 Baseline (7 days): number analyzed (Participants) | 0 | 1
  Subject 11 Baseline (7 days) |  | 4
  Subject 11 28-day period 4 (15 days): number analyzed (Participants) | 0 | 1
  Subject 11 28-day period 4 (15 days) |  | 0
  Subject 12 Baseline (4 days): number analyzed (Participants) | 1 | 0
  Subject 12 Baseline (4 days) | NA — Data were collected on 4 days, therefore the baseline value was not valid |
  Subject 12 28-day period 1 (27 days): number analyzed (Participants) | 1 | 0
  Subject 12 28-day period 1 (27 days) | 18.667 |
  Subject 13 Baseline (7 days): number analyzed (Participants) | 0 | 1
  Subject 13 Baseline (7 days) |  | 8
  Subject 13 28-day period 4 (21 days): number analyzed (Participants) | 0 | 1
  Subject 13 28-day period 4 (21 days) |  | 1.333
  Subject 14 Baseline (3 days): number analyzed (Participants) | 1 | 0
  Subject 14 Baseline (3 days) | NA — Data were collected on 3 days, therefore the baseline value was not valid |
  Subject 14 28-day period 3 (10 days): number analyzed (Participants) | 1 | 0
  Subject 14 28-day period 3 (10 days) | 0 |

7. Secondary Outcome: Number of MHD Responders (Defined as a ≥50% Reduction in MHD)
Description: A subject was considered a responder if they had at least a 50% reduction in MHD from baseline to Week 24. Subjects who dropped out prior to Week 24 were considered non-responders.
Time Frame: Baseline to Week 24
Population: The number of responders is provided for all subjects (including those who were considered non-responders because they dropped out of the study prior to Week 24) and for subjects who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 8 | 6
Participants
  Number of responders (subjects who completed the study): number analyzed (Participants) | 3 | 1
  Number of responders (subjects who completed the study) | 1 | 0
  Number of responders (all subjects) | 1 | 0

8. Secondary Outcome: Number of Moderate to Severe MHD Responders (Defined as a ≥50% Reduction in Moderate to Severe MHD)
Description: A subject was considered a responder if they had at least a 50% reduction in moderate to severe MHD from baseline to Week 24. Subjects who dropped out prior to Week 24 were considered non-responders.
Time Frame: Baseline to Week 24
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 8 | 6
Participants
  Number of responders (subjects who completed the study): number analyzed (Participants) | 3 | 1
  Number of responders (subjects who completed the study) | 2 | 0
  Number of responders (all subjects) | 2 | 0

9. Secondary Outcome: Headache Severity
Description: Headache severity was assessed by a 10-point Numeric Rating Scale (NRS), 0-10 where 0 = no pain and 10 = most severe pain. Severity of headaches was assessed on days where a headache occurred. Headache free days were not counted. Baseline headache severity was calculated over the 7 days prior to the randomization visit; at least 5 of 7 days of headache severity data had to be recorded by the subject to obtain a valid baseline value.
  * 28-day period 1 = Weeks 1-4
  * 28-day period 2 = Weeks 5-8
  * 28-day period 3 = Weeks 9-12
  * 28-day period 4 = Weeks 13-16
  * 28-day period 5 = Weeks 17-20
  * 28-day period 6 = Weeks 21-24
Time Frame: Baseline to Week 24
Population: Data presented represents collected data from individual subjects. For anonymity, study-assigned subject IDs are not included and subject numbers used throughout ClinicalTrials.gov results do not consistently relate to the same subjects.
  Number of days on which severity data were collected for each subject during the 7-day baseline and the last 28-day periods are provided in row titles.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 8 | 6
score on a scale
  Subject 1 baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 1 baseline (5 days) | 6 [4 to 7] |
  Subject 1 28-day period 6 (14 days): number analyzed (Participants) | 1 | 0
  Subject 1 28-day period 6 (14 days) | 4 [2 to 7] |
  Subject 2 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 2 Baseline (5 days) | 3 [2 to 4] |
  Subject 2 28-day period 6 (3 days): number analyzed (Participants) | 1 | 0
  Subject 2 28-day period 6 (3 days) | 4 [2 to 6] |
  Subject 3 Baseline (7 days): number analyzed (Participants) | 0 | 1
  Subject 3 Baseline (7 days) |  | 4 [2 to 5]
  Subject 3 28-day period 6 (9 days): number analyzed (Participants) | 0 | 1
  Subject 3 28-day period 6 (9 days) |  | 8 [3 to 8]
  Subject 4 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 4 Baseline (5 days) | 5 [3 to 7] |
  Subject 4 28-day period 4 (11 days): number analyzed (Participants) | 1 | 0
  Subject 4 28-day period 4 (11 days) | 7 [6 to 8] |
  Subject 5 Baseline (1 day): number analyzed (Participants) | 1 | 0
  Subject 5 Baseline (1 day) | NA [NA to NA] — Data were collected on 1 day, therefore the baseline value was not valid |
  Subject 5 28-day period 4 (2 days): number analyzed (Participants) | 1 | 0
  Subject 5 28-day period 4 (2 days) | 3 [3 to 3] |
  Subject 6 Baseline (3 days): number analyzed (Participants) | 0 | 1
  Subject 6 Baseline (3 days) |  | NA [NA to NA] — Data were collected on 3 days, therefore the baseline value was not valid
  Subject 6 28-day period 2 (5 days): number analyzed (Participants) | 0 | 1
  Subject 6 28-day period 2 (5 days) |  | 2 [2 to 9]
  Subject 7 Baseline (0 days): number analyzed (Participants) | 0 | 0
  Subject 7 28-day period 4 (4 days): number analyzed (Participants) | 0 | 1
  Subject 7 28-day period 4 (4 days) |  | 2 [2 to 2]
  Subject 8 Baseline (6 days): number analyzed (Participants) | 0 | 1
  Subject 8 Baseline (6 days) |  | 4.5 [3 to 6]
  Subject 8 28-day period 2 (8 days): number analyzed (Participants) | 0 | 1
  Subject 8 28-day period 2 (8 days) |  | 7 [6 to 9]
  Subject 9 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 9 Baseline (5 days) | 4 [3 to 8] |
  Subject 9 28-day period 6 (11 days): number analyzed (Participants) | 1 | 0
  Subject 9 28-day period 6 (11 days) | 1 [1 to 2] |
  Subject 10 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 10 Baseline (5 days) | 7 [7 to 8] |
  Subject 10 28-day period 4 (8 days): number analyzed (Participants) | 1 | 0
  Subject 10 28-day period 4 (8 days) | 6 [3 to 7] |
  Subject 11 Baseline (5 days): number analyzed (Participants) | 0 | 1
  Subject 11 Baseline (5 days) |  | 5 [4 to 8]
  Subject 11 28-day period 4 (3 days): number analyzed (Participants) | 0 | 1
  Subject 11 28-day period 4 (3 days) |  | 4 [2 to 4]
  Subject 12 Baseline (4 days): number analyzed (Participants) | 1 | 0
  Subject 12 Baseline (4 days) | NA [NA to NA] — Data were collected on 4 days, therefore the baseline value was not valid |
  Subject 12 28-day period 1 (25 days): number analyzed (Participants) | 1 | 0
  Subject 12 28-day period 1 (25 days) | 6 [3 to 9] |
  Subject 13 Baseline (6 days): number analyzed (Participants) | 0 | 1
  Subject 13 Baseline (6 days) |  | 4.5 [3 to 7]
  Subject 13 28-day period 4 (2 days): number analyzed (Participants) | 0 | 1
  Subject 13 28-day period 4 (2 days) |  | 4 [3 to 5]
  Subject 14 Baseline (0 days): number analyzed (Participants) | 0 | 0
  Subject 14 28-day period 3 (1 day): number analyzed (Participants) | 1 | 0
  Subject 14 28-day period 3 (1 day) | 3 [3 to 3] |

10. Secondary Outcome: Use of Acute Headache Analgesic Medications (Acute Headache Analgesics in Days Per Month)
Description: Number of days recorded in a 28-day window, where at least one dose of an acute headache analgesic was recorded.
  The baseline acute headache analgesic use was calculated over the 7 days prior to the randomization visit; at least 5 of 7 days had to be recorded by the subject to obtain a valid baseline value.
  The number of acute headache analgesic use days was linearly scaled for each subject to give the number of acute headache analgesic use days during the baseline period and the last 28-day period during which headache data were collected on more than 7 days for each subject prior to study completion or discontinuation.
  * 28-day period 1 = Weeks 1-4
  * 28-day period 2 = Weeks 5-8
  * 28-day period 3 = Weeks 9-12
  * 28-day period 4 = Weeks 13-16
  * 28-day period 5 = Weeks 17-20
  * 28-day period 6 = Weeks 21-24
Time Frame: Baseline to Week 24
Population: Data presented represents collected data from individual subjects. For anonymity, study-assigned subject IDs are not included here, and subject numbers used throughout the ClinicalTrials.gov results do not consistently relate to the same subjects. The number of days on which analgesic use were collected for each subject during the 7-day baseline and the last 28-day periods are provided in parentheses in row titles.
Measure: Number; unit: Acute headache analgesics days per month
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 8 | 6
Acute headache analgesics days per month
  Subject 1 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 1 Baseline (5 days) | 0 |
  Subject 1 28-day period 6 (14 days): number analyzed (Participants) | 1 | 0
  Subject 1 28-day period 6 (14 days) | 6 |
  Subject 2 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 2 Baseline (5 days) | 16.8 |
  Subject 2 28-day period 6 (3 days): number analyzed (Participants) | 1 | 0
  Subject 2 28-day period 6 (3 days) | 0 |
  Subject 3 Baseline (7 days): number analyzed (Participants) | 0 | 1
  Subject 3 Baseline (7 days) |  | 4
  Subject 3 28-day period 6 (9 days): number analyzed (Participants) | 0 | 1
  Subject 3 28-day period 6 (9 days) |  | 24.89
  Subject 4 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 4 Baseline (5 days) | 0 |
  Subject 4 28-day period 4 (11 days): number analyzed (Participants) | 1 | 0
  Subject 4 28-day period 4 (11 days) | 0 |
  Subject 5 Baseline (1 day): number analyzed (Participants) | 1 | 0
  Subject 5 Baseline (1 day) | NA — Data were collected on 1 day, therefore the baseline value was not valid |
  Subject 5 28-day period 4 (2 days): number analyzed (Participants) | 1 | 0
  Subject 5 28-day period 4 (2 days) | 0 |
  Subject 6 Baseline (3 days): number analyzed (Participants) | 0 | 1
  Subject 6 Baseline (3 days) |  | NA — Data were collected on 3 days, therefore the baseline value was not valid
  Subject 6 28-day period 2 (5 days): number analyzed (Participants) | 0 | 1
  Subject 6 28-day period 2 (5 days) |  | 11.2
  Subject 7 Baseline (0 days): number analyzed (Participants) | 0 | 0
  Subject 7 28-day period 4 (4 days): number analyzed (Participants) | 0 | 1
  Subject 7 28-day period 4 (4 days) |  | 0
  Subject 8 Baseline (6 days): number analyzed (Participants) | 0 | 1
  Subject 8 Baseline (6 days) |  | 0
  Subject 8 28-day period 2 (8 days): number analyzed (Participants) | 0 | 1
  Subject 8 28-day period 2 (8 days) |  | 10.5
  Subject 9 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 9 Baseline (5 days) | 16.8 |
  Subject 9 28-day period 6 (11 days): number analyzed (Participants) | 1 | 0
  Subject 9 28-day period 6 (11 days) | 0 |
  Subject 10 Baseline (5 days): number analyzed (Participants) | 1 | 0
  Subject 10 Baseline (5 days) | 11.2 |
  Subject 10 28-day period 4 (8 days): number analyzed (Participants) | 1 | 0
  Subject 10 28-day period 4 (8 days) | 14 |
  Subject 11 Baseline (5 days): number analyzed (Participants) | 0 | 1
  Subject 11 Baseline (5 days) |  | 5.6
  Subject 11 28-day period 4 (3 days): number analyzed (Participants) | 0 | 1
  Subject 11 28-day period 4 (3 days) |  | 0
  Subject 12 Baseline (4 days): number analyzed (Participants) | 1 | 0
  Subject 12 Baseline (4 days) | NA — Data were collected on 4 days, therefore the baseline value was not valid |
  Subject 12 28-day period 1 (25 days): number analyzed (Participants) | 1 | 0
  Subject 12 28-day period 1 (25 days) | 13.44 |
  Subject 13 Baseline (6 days): number analyzed (Participants) | 0 | 1
  Subject 13 Baseline (6 days) |  | 9.333
  Subject 13 28-day period 4 (2 days): number analyzed (Participants) | 0 | 1
  Subject 13 28-day period 4 (2 days) |  | 14
  Subject 14 Baseline (0 days): number analyzed (Participants) | 0 | 0
  Subject 14 28-day period 3 (1 day): number analyzed (Participants) | 1 | 0
  Subject 14 28-day period 3 (1 day) | 0 |

11. Secondary Outcome: Visual Acuity
Description: Corrected visual acuity will be recorded using a Logarithm of the Minimum Angle of Resolution (LogMAR) scoring chart, with a range of -0.3 to 1.00, where a lower score indicates better visual acuity.
Time Frame: Baseline to Week 24
Population: Data were not collected from subjects with qualifying study eyes for this endpoint.
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Patients With Treatment Failure
Description: Treatment failure is defined as the initiation of either medical therapy or a surgical intervention to lower ICP during the study.
Time Frame: Baseline to Week 24
Measure: Number; unit: participants
Arm/Group | Presendin | Placebo
Number analyzed (Participants) | 8 | 6
participants
  Treatment failure suspected | 0 | 1
  Treatment failure confirmed | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of up to 30 weeks, from the signing of the informed consent form to the end of the follow-up period.
Description: Adverse events reported from the signing of the informed consent form to the start of dosing of the drug product (active or placebo) are reported for the "All subjects pre-treatment group". Treatment-emergent adverse events (adverse events with an onset after the start of dosing of the drug product [active or placebo] or an event with an onset before dosing but that worsened in severity after the start of dosing) are reported for the "Placebo" and "Presendin" groups.
Groups:
- All Subjects Pre-treatment: All subjects after signing the informed consent form and before being assigned to treatment groups or the start of dosing of the drug product
Arm/Group | Presendin | Placebo | All Subjects Pre-treatment
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/14
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Presendin (N=8) | Placebo (N=6) | All Subjects Pre-treatment (N=14)
Injection site mass (General disorders) | 2 (2) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site hypersensitivity (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site indentation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) — Injection site reaction due to demonstration kit

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, planned analyses were not fully conducted but were restricted to the most relevant safety endpoints as per the abbreviated SAP v1. Outcome measure (efficacy) data are raw data from individual subjects, with minimal analysis; e.g., where an outcome measure specified change from baseline to Week 24, baseline and Week 24 values are presented. Efficacy data were not subject to the same verification as safety data and no efficacy conclusions should be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Investigator wishes to publish anything related to the trial, then they must provide the Sponsor with the draft publication and allow them no less than 30 days to review the document. The Investigator cannot publish without written authorisation from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT05347147/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT05347147/SAP_001.pdf